CLINICAL TRIAL: NCT00671476
Title: Intraductal Therapy of DCIS: A Presurgery Study
Brief Title: Doxorubicin Hydrochloride Liposome in Treating Women With Ductal Carcinoma in Situ Undergoing Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Susan Love Research Foundation (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: CDR0000594671; DSLRF-SJHCA-00003154; SJHCA-00003154
Record Dates: First submitted 2008-05-02; First posted 2008-05-05 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — DNA Methylation; In Situ Hybridization, Fluorescence; Polymerase Chain Reaction; Immunoenzyme Techniques; Immunohistochemistry; Neoadjuvant Therapy

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride
Genetic: DNA methylation analysis
Genetic: TdT-mediated dUTP nick end labeling assay
Genetic: fluorescence in situ hybridization
Genetic: loss of heterozygosity analysis
Genetic: polymerase chain reaction
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: breast duct lavage
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This clinical trial is studying the side effects of doxorubicin hydrochloride liposome and to see how well it works in treating women with ductal carcinoma in situ undergoing surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To demonstrate the efficacy and safety of neoadjuvant intraductal pegylated liposomal doxorubicin hydrochloride in women with ductal breast carcinoma in situ undergoing surgery.
* To demonstrate the ability to identify and cannulate the duct demonstrating precancerous disease in these women.
* To integrate the Humboldt Community Breast Health Project into the planning and execution of this study.

OUTLINE: Patients undergo identification of the intraductal lesions via cannulization. Patients receive pegylated liposomal doxorubicin hydrochloride (PLD) intraductally through the inserted cannula. Some patients are randomized to receive saline instead of PLD. Within 4-6 weeks, all patients undergo surgery.

Patients undergo tissue and ductal fluid sample collection at baseline and at surgery for correlative laboratory studies. Tissue samples are assessed for histomorphology, proliferation (Ki67), cell death (apoptosis index), genetic markers, necrosis, inflammation, and loss of heterozygosity by HE stain, IHC, TUNEL, and PCR. Nipple aspirate and ductal lavage fluid samples are analyzed for cytomorphology (cellular atypia), proliferation (Ki67), cell death (TUNEL), differentiation (G-actin), and genetic markers (FISH) by quantitative fluorescence image analysis. Samples are also analyzed for bFGF and CEA by ELISA, and methylation by PCR.

After completion of study therapy, patients are followed every 6 months for at least 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ductal breast carcinoma in situ by core needle biopsy

  * No pathological invasive or microinvasive disease in the affected breast
* Mammographic microcalcifications are limited to one ductal system or one quadrant of breast
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Must be able to undergo necessary surgery
* Not pregnant

PRIOR CONCURRENT THERAPY:

* No prior surgery or radiotherapy to the recently diagnosed breast
* More than 12 months since prior chemotherapy
* No prior subareolar breast surgery to the affected breast
* Not concurrently involved in a research protocol for unapproved new drug evaluation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy
Safety
Ability to identify and cannulate the duct
Integration of the Humboldt Community Breast Health Project into the planning and execution of this study

CONTACTS AND LOCATIONS:
Overall Officials: Susan Love, MD, MBA, Principal Investigator — Dr. Susan Love Research Foundation
Locations (2):
- United States (2):
  - St. Joseph Hospital, Eureka, California
  - Doctor Susan Love Research Foundation, Santa Monica, California